CLINICAL TRIAL: NCT02594358
Title: Caffeine in Amblyopia Study
Acronym: CAS
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Could not recruit
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Michael Repka, Professor of Ophthalmology, Johns Hopkins University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00066787
Record Dates: First submitted 2015-10-30; First posted 2015-11-03 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Amblyopia
Keywords: Caffeine
MeSH Terms: conditions — Amblyopia | interventions — Caffeine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caffeine 20 mg (Active Comparator): Patching plus once daily caffeine for 12 weeks
  Interventions: Drug: Caffeine
- Caffeine 40 mg (Active Comparator): Patching plus once daily caffeine for 12 weeks
  Interventions: Drug: Caffeine

INTERVENTIONS:
Drug: Caffeine — 20 MG OR 40 MG ONCE DAILY ALONG WITH PATCHING

SUMMARY:
Prospective data on the visual acuity response in children treated by patching concurrently treated with caffeine and estimate the magnitude of effect that might be seen in a randomized trial (if no improvement in acuity is seen, this would be sufficient evidence to decide not to conduct a randomized, double blind trial).

Collect prospective data on the tolerability of caffeine in two dosages as an adjuvant treatment for amblyopia and provide limited data on its safety.

Evaluate the potential for a dietary intervention to enhance the acceptance and tolerability of patching on the child and family.

Demonstrate recruitment potential of subjects to participate in a dietary intervention study.

ELIGIBILITY:
Inclusion Criteria:

* Amblyopia from strabismus and amblyopia

Exclusion Criteria:

* Known intolerance to caffeine
* Diagnosis and/or treatment of attention deficit/hyperactivity disorder
* Presence of an ocular cause for reduced visual acuity
* Myopia with a special equivalent -6.00 diopters
* Current vision therapy or orthoptics - any type
* Ocular cause for reduced visual acuity
* Prior intraocular or refractive surgery
* History of narrow-angle glaucoma
* Strabismus surgery planned within 16 weeks
* Nystagmus per se does not exclude the subject if the above visual acuity criteria are met
* Known skin reactions to patch or bandage adhesives
* Known allergy or intolerance to food dyes
* Current treatment with topical atropine eyedrops
* Menarche, pregnancy or lactation
* Use of any of the following medications which may affect caffeine metabolism: nafcillin, verapamil, fluvoxamine, ciprofloxacin and other fluoroquinolones, modafinil, nafcillin, and omeprazole

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 12 weeks
  Quantitative improvement in high resolution visual acuity measured at 3 meters

SECONDARY OUTCOMES:
Questionnaire | 12 weeks
  A multiquestion survey is adminsitered to the subjects specifically asking about side effects and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Michael X Repka, MD, MBA, Study Chair — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States